CLINICAL TRIAL: NCT03224442
Title: Clinical Evaluation of Peri-Implant Soft Tissue Around Immediately Placed Implants Using PRF Membrane Versus The Palatal Pedicle Soft Tissue Graft: A Randomized Controlled Clinical Trial.
Brief Title: Soft Tissue Evaluation Around Implants Using Prf or a Palatal Pedicle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Andrew George Edward Aziz, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Philoprotocol
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Soft Tissue Augmentation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF with immediate implants (Experimental): Immediate implants placed and covered with two prf layers
  Interventions: Procedure: PRF
- palatal pedicle graft (Active Comparator): immediate implant placement followed by soft tissue augmentation by oalatal pedicle graft
  Interventions: Procedure: Palatal Pedicle

INTERVENTIONS:
Procedure: PRF — soft tissue augmentation by prf
  Arms: PRF with immediate implants
Procedure: Palatal Pedicle — soft tissue augmentation by palatal pedicle
  Arms: palatal pedicle graft

SUMMARY:
Clinical Evaluation of Peri-Implant Soft Tissue Around Immediately Placed Implants Using PRF Membrane Versus The Palatal Pedicle Soft Tissue Graft: A Randomized Controlled Clinical Trial.

DETAILED DESCRIPTION:
Immediate implant will be place and followed by soft tissue augmentation by PRF or palatal pedicle and the primary outcome is the pink esthetic score

ELIGIBILITY:
Inclusion criteria

1. Absence of periodontal disease or a periapical infection
2. Adequate native bone to achieve implant primary stability
3. The need for a single-tooth replacement in the anterior maxilla (from the second bicuspid to the second bicuspid), subsequent to an inevitable tooth extraction.

Exclusion criteria

1. Systemic conditions/disease that contraindicated surgery
2. Radiation therapy in the head and neck region or chemotherapy during the 12 months prior to surgery.
3. Patients who have any habits that might jeopardize the osseointegration process, such as current smokers.
4. Patients with parafunctional habits that produce overload on implant, such as bruxism and clenching.
5. Patients who have inadequate interarch space for the prosthetic part.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score | 5 months
  photographs

SECONDARY OUTCOMES:
facial gingival thickness | 5 months
  probe
mid-buccal gingival level | 5 months
  probe
interproximal gingival level | 5 months
  probe
- width of keratinized gingiva (KG | 5 months
  probe
Crestal bone loss | 5 months
  CBCT
Implant stability | 5 months
  ostel
Pain | 5 months
  VAS